CLINICAL TRIAL: NCT06785584
Title: Efficacy and Safety of Ensartinib in Neoadjuvant Therapy for Stage IIA - IIIB (Operable or Potentially Operable) ALK-Positive Lung Adenocarcinoma ：A Multicenter, Real-World Clinical Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024ENT01
Record Dates: First submitted 2024-11-26; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-11

CONDITIONS: ALK-positive Advanced NSCLC; ALK-positive Non-small Cell Lung Cancer (NSCLC); MPR; Neoadjuvant Therapy
Keywords: Ensartinib; Neoadjuvant Therapy; ALK-Positive Lung Adenocarcinoma; MPR
MeSH Terms: interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ensartinib For Neoadjuvant Therapy (Experimental): receive neoadjuvant treatment with ensartinib 225 mg once a day, po. for 2 consecutive cycles (56 days) to evaluate possibility of surgery, or discontinue the treatment because of disease recurrence or intolerable toxicity
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — receive neoadjuvant treatment with ensartinib 225 mg once a day, po. for 2 consecutive cycles (56 days) to evaluate possibility of surgery, or discontinue the treatment because of disease recurrence or intolerable toxicity

SUMMARY:
According to the Global Cancer Statistics 2022 report, lung cancer is the most common type of cancer (12.4% of the total) and the leading cause of cancer deaths (18.7% of total cancer deaths). According to the pathological classification of patients, lung cancer is divided into small cell lung cancer and non-small cell lung cancer, of which non-small cell lung cancer (NSCLC) accounts for 80-85% of all lung cancer.

Surgery is the preferred treatment for patients with early-stage lung cancer, according to the 2024 CSCO Guidelines. However, most patients have the possibility of recurrence and metastasis after surgery. The 5-year survival rate of patients with stage IA NSCLC is 80%-90%, but the 5-year survival rate of patients with stage ⅢB NSCLC drops to 40%. Neoadjuvant therapy has become an important part of the treatment of non-small cell lung cancer (NSCLC) in order to prolong the survival of patients.

In the past few years, many driver genes of NSCLC have been identified, and anaplastic lymphoma kinase (ALK) is one of them. ALK was first identified in anaplastic large cell lymphoma (ALCL). Studies at home and abroad have shown that ALK-rearranged (positive)NSCLC accounts for about 3%-7% of all NSCLC patients.

Many studies have suggested that ALK-TKI is clinically feasible as a neoadjuvant therapy for ALK positve patients with locally advanced NSCLC.

The investigators designed this study to explore the efficacy of enshatinib neoadjuvant therapy in patients with stage IIA to III ALK-positive lung adenocarcinoma

DETAILED DESCRIPTION:
According to the Global Cancer Statistics 2022 report, lung cancer is the most common type of cancer (12.4% of the total) and the leading cause of cancer deaths (18.7% of total cancer deaths). The statistics of the National Cancer Center of China shows that there are about 1 061 thousand new cases and 733 thousand deaths of lung cancer in China every year, which account for the first incidence and mortality of malignant tumors in China. According to the pathological classification of patients, lung cancer is divided into small cell lung cancer and non-small cell lung cancer, of which non-small cell lung cancer (NSCLC) accounts for 80-85% of all lung cancer.

Surgery is the preferred treatment for patients with early-stage lung cancer, according to the 2024 CSCO Guidelines. However, most patients have the possibility of recurrence and metastasis after surgery. The 5-year survival rate of patients with stage IA NSCLC is 80%-90%, but the 5-year survival rate of patients with stage ⅢB NSCLC drops to 40%. Neoadjuvant therapy has become an important part of the treatment of non-small cell lung cancer (NSCLC) in order to prolong the survival of patients.

In the past few years, many driver genes of NSCLC have been identified, and anaplastic lymphoma kinase (ALK) is one of them. ALK was first identified in anaplastic large cell lymphoma (ALCL). Studies at home and abroad have shown that ALK-rearranged (positive)NSCLC accounts for about 3%-7% of all NSCLC patients.

Many studies such as The SAKULA study,The ALNEO Study have suggested that ALK-TKI is clinically feasible as a neoadjuvant therapy for ALK positve patients with locally advanced NSCLC.

Ensartinib is a novel potent and highly selective second-generation ALK inhibitor, which has a good selective inhibition effect on c-Met. Structurally, Ensartinib is similar to crizotinib, but Ensartinib has stronger binding to ALK and better selectivity than crizotinib, and both in vitro and in vivo experiments have shown the potential of ensartinib for crizotinib-resistant tumors.

The safety profile of ensartinib was manageable. In the eXalt3 study, the most common adverse events of all grades in the ensartinib group were rash, pruritus, and elevated aminotransferase (ALT, AST).

The eXalt3 study confirmed that first-line use of ensartinib can significantly improve mPFS compared with crizotinib in ALK-positive NSCLC patients, and ensartinib provides better efficacy and safety, making it a new first-line treatment option for ALK-positive NSCLC patients.

ALK inhibitors have brought great survival benefits to ALK-positive advanced NSCLC, but the exploration of ALK inhibitors in early-stage patients has just begun,with no authoritative results have been published. TThe investigators designed this study to explore the efficacy of neoadjuvant treatment with ensartinib in patients with stage IIA-IIB ALK-positive lung adenocarcinoma who had undergone neoadjuvant chemotherapy for ALK mutation.

The primary goal of this study is to evaluate the major pathological response (MPR) to neoadjuvant ensartinib in patients with resectable stage IIA to IIIb ALK-positive non-small cell lung cancer (NSCLC).

The secondary objectives are to evaluate the complete pathological response (pCR), objective response rate (ORR), and safety of neoadjuvant ensartinib in patients with resectable stage IIA-IIIb ALK-positive non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Histologically or cytologically confirmed lung adenocarcinoma
* Evaluated resectable TNM stage IIA-IIIB (operable or potentially operable) non-small cell lung cancer (NSCLC)
* Alk-positive as determined by immunohistochemistry (IHC), fluorescence in situ hybridization (FISH), next-generation sequencing (NGS), or other non-specific sequencing methods，before treatment with ALK inhibitors
* Measurable lesions were determined with the use of the Response Evaluation Criteria in Solid Tumors (RECIST 1.1 criteria) on CT scans
* Magnetic resonance imaging (MRI) or CT scans of the brain show no metastatic disease
* Tumors contained components of squamous cell carcinoma, large-cell neuroendocrine carcinoma, or small-cell carcinoma
* Severe infections, including COVID-19, including but not limited to hospitalization due to complications of infection within the 4 weeks prior to starting study treatment
* Have not received chemotherapy, radiotherapy, or biological therapy
* Hemoglobin ≥100 g/L(which can be maintained or exceeded by blood transfusion); Absolute neutrophil count ≥2.0×109/L; Platelet count ≥100×109/L
* Total bilirubin ≤1.5 times upper limit of normal; ALT and AST≤2.5 times the upper limit of normal; CREA ≤1.5 times the upper limit of normal and CREA clearance ≥60mL/min
* Women of childbearing age (15 to 49 years) must undergo a urine pregnancy test within 7 days before starting treatment and the result is negative
* Informed consent is obtained from patients or their legal representatives
* Able to swallow oral medications normally
* ECOG behavior status score is 0 to 1
* Men and women of reproductive age agree to use a reliable method of contraception before entering the trial, during the study and up to eight weeks after discontinuation
* Stable health status, including no acute exacerbations of chronic diseases, serious infections, or major surgeries during the first 4 weeks of enrollment, as indicated in other inclusion/exclusion criteria

Exclusion Criteria:

* Have received any systemic anti-cancer treatment for locally advanced non-small cell lung cancer, including chemotherapy, biotherapy (including ALK-TKI), immunotherapy, or any investigational drug
* PET-CT scan or biopsy results showing unresectable stage III and IV disease with distant metastasis (including malignant pleural effusion)
* Patients who had a cancer other than NSCLC within 5 years before the initiation of study treatment
* Allergy to ensartinib or any of the ingredients in this product
* Previous history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonia requiring hormone therapy, or any clinically proven active interstitial lung disease;Baseline CT scans found idiopathic pulmonary fibrosis
* Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow preparations, or previous major bowel resection resulting in inadequate absorption of ensartinib
* Any unstable systemic illness, including active infection, uncontrolled hypertension, unstable angina, angina with onset within the last 3 months, congestive heart failure (≥ New York Heart Association [NYHA] class II), myocardial infarction (within 6 months before enrollment), severe arrhythmias requiring medical therapy, or hepatic, renal, or metabolic disease
* Human immunodeficiency virus (HIV) infection
* Pregnant or lactating women
* A definite past history of neurological or psychiatric disorders, including epilepsy or dementia
* History of organ transplantation
* Rheumatic immune-related diseases
* Other cases that the researcher deemed unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate(MPR) | From enrollment to the end of treatment at 8 weeks
  The proportion of patients with ≤10% residual viable tumor cells in the resected primary tumor and metastatic lymph nodes after completion of neoadjuvant therapy

SECONDARY OUTCOMES:
Pathological complete response rate (pCR) | From enrollment to the end of treatment at 8 weeks
  Proportion of patients who had no residual tumor in the resected primary tumor and metastatic lymph nodes after completion of neoadjuvant therapy
Objective Response Rate (ORR) | From enrollment to the end of treatment at 8 weeks
  The proportion of patients with a complete response (CR) or partial response (PR) among all patients, as assessed according to RECIST, version 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes